CLINICAL TRIAL: NCT01345552
Title: Phase II Study of Stereotactic Radiosurgery for Patients With Oligo-recurrent Disease
Brief Title: Radiosurgery for Patients Recurrent Oligometastatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Burton (Other)
Responsible Party: Sponsor-Investigator, Steven Burton, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 10-028
Record Dates: First submitted 2011-02-24; First posted 2011-05-02 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Oligometastatic Disease
Keywords: Oligo mets; Oligometastatic disease; Stereotactic Body Radiotherapy (SBRT) (Stereotactic radiosurgery (SRS) plus stereotactic radiotherapy (SRT))
MeSH Terms: conditions — Snyder Robinson syndrome | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SBRT (Other)
  Interventions: Radiation: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (SRS) — Dose and fractionation will be dependent on the lesion location and lesion size and is up to the exact fractionation and dose is at the discretion of the treating physician. A minimum of 48 hours must be used in between SRS treatments at each site. Note that patients can have SRS everyday or multiple SRS sessions in one day as long as the minimum time for each treatment site is met. For example, if two lung lesions, brain, adrenal, and liver sites were being treated both lung sites could be treated Monday, Wednesday, and Friday and the adrenal, liver and brain lesions treated Tuesday, Thursday
  Other Names: CyberKnife; Trilogy; True Beam

SUMMARY:
This study will evaluate the feasibility of radiosurgery for all metastatic sites in patients presenting with oligometastatic disease, defined here as 5 or fewer sites of metastatic disease involving 3 or fewer organ systems.

DETAILED DESCRIPTION:
Death from metastatic cancer is a common cause of death, accounting for 80-90% of cancer deaths. The classic thought process is that metastatic disease represents the continuum such that known metastatic disease is an inevitable harbinger for subsequent metastatic disease. However, it has been reported that a subset of patients with limited volume metastatic disease may have a better prognosis if given aggressive therapy. This group of patients has become known as "oligometastatic". These patients are potentially curable with stereotactic radiosurgery (SRS) or stereotactic radiotherapy (SRT) (collectively referred to as stereotactic body radiotherapy or SBRT) to the metastatic disease sites in combination with standard curative therapy to the primary site. Patients in this study receive SRS/SBRT to all sites of oligometastatic disease.

ELIGIBILITY:
Inclusion Criteria:

3.1 Conditions for Patient Eligibility

3.1.1 Pathologically (histologically or cytologically) proven diagnosis of solid malignancy 3.1.2 Eligible disease sites include the following

* Breast
* Prostate
* GI (including colorectal, anal, esophagus, pancreas, gastric with the exception of patients with colon cancer and liver-only metastatic disease )
* Head and neck
* Skin (melanoma and squamous cell carcinoma)
* Lung (both small cell and non-small cell)
* Sarcoma (both soft tissue and bone)
* Gynecologic (endometrial, cervical, ovarian, vaginal, vulvar)

3.1.3 Patients are stage IV (M1) or recurrent with any combination of T and N with oligometastatic disease as defined by 5 or fewer total sites of metastatic disease 3.1.4 Can have recurrent disease from the primary disease (this is definition of oligorecurrent disease) but cannot have any other primary cancer diagnosed or treated within the last 3 years other than cutaneous skin cancer.

3.1.5 Prior systemic chemotherapy is allowable 3.1.4 Zubrod Performance Status 0-1 3.1.5 Age ≥ 18 3.1.6 CBC/differential obtained within 4 weeks prior to registration on study, with adequate bone marrow function defined as follows: 3.1.6.1 Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3; 3.1.6.2 Platelets ≥ 100,000 cells/mm3; 3.1.6.3 Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.); 3.1.7 Women of childbearing potential and male participants must practice adequate contraception 3.1.8 Patient must provide study specific informed consent prior to study entry

Exclusion Criteria:

3.2.1 Ineligible disease sites include the following

* Lymphoma
* Leukemia
* Multiple myeloma
* Primary CNS
* Peritoneal carcinomatosis
* Colon cancer with liver-only metastatic disease that is treatable with surgical resection 3.2.2 Other
* Diffuse metastatic spread confined to one organ system is ineligible; examples of this include leptomeningeal spread in the CNS and peritoneal carcinomatosis.
* Metastatic disease sites must be treatable with stereotactic radiosurgery (at discretion of treating physician). Patients with oligometastatic sites not amenable to SRS treatment, either through size or locations, are ineligible for this trial.

3.2.4 Severe, active co-morbidity, defined as follows: 3.2.4.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; 3.2.4.2 Transmural myocardial infarction within the last 6 months; 3.2.4.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; 3.2.4.4 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.

3.2.5 Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

3.2.6 Patients unable to have an FDG-PET scan, either through insurance coverage, patient decision or other reason are not eligible for this study.

3.2.7 Oligometastatic disease sites not eligible based on concern for toxicity:

* trachea involvement (direct invasion, tumors close to or abutting trachea are eligible)
* heart (direct invasion or involvement, pericardial lymph nodes can be treated) 3.2.8 Patients unable to have SRS through insurance coverage or ability to pay for SRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events Related to Treatment | Up to 5 years
  Adverse Events as measured by CTCAE version 4.0, possibly, probably or definitely related to study treatment.

SECONDARY OUTCOMES:
Serious Adverse Events related to treatment | Up to 5 years
  Serious Adverse Events as measured by CTCAE version 4.0, possibly, probably or definitely related to study treatment.
The Functional Assessment of Cancer Therapy - General (FACT-G) | 5 years
  A a self-administered, 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Scaling of items: Five-point scale from 0 (not at all) to 4 (very much). Scoring: Subscale scores added to obtain total score. Alternative scoring includes the Trial Outcome Index (TOI), which is the sum of the Physical, Functional, Cancer Subscales. The TOI is reported to be an efficient and precise summary index of physical and functional outcomes. Higher scores indicated better quality of life.
Local control of metastatic sites | Up to 5 years
  Proportion of patients with local control is defined as stable disease (SD), partial response (PR), or complete response (CR) in the target lesion, per RECIST v1.1. Complete Response (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Overall survival (OS) | Up to 5 years
  The (median) length of time from enrollment to confirmed death from any cause.
Analysis of patterns of failure post-SRS/SBRT | Up to 5 years
  Proportion of patients with local failure (progressive disease (PD) within the target lesion. Per RECIST v1.1: Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burton, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center - Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No